CLINICAL TRIAL: NCT05327504
Title: Written Exposure Therapy (WET) as a Brief Trauma Treatment for Veterans With Co-occurring Substance Use Disorders and PTSD
Brief Title: Written Exposure Therapy for Veterans With SUD and PTSD
Acronym: WET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBP-010-21F
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Substance Use Disorders; Posttraumatic Stress Disorder
Keywords: Addiction; Trauma and Stress Related Disorders; Substance Use Disorder; PTSD; Comorbidity
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic; Behavior, Addictive; Trauma and Stressor Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial within a Substance Use Disorder (SUD) clinic to evaluate whether treatment as usual (TAU) plus Written Exposure Therapy (WET) is superior to TAU augmented by a neutral topic writing on both PTSD and addiction outcomes for Veterans who present to SUD treatment with comorbid SUD/PTSD.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to randomization status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Written Exposure Therapy (Experimental): Written Exposure Therapy (WET) plus Treatment As Usual (TAU). WET is a 5 session, evidence-based trauma-focused written narrative exposure treatment. At each session, patients are instructed to write about the same trauma event and therapists provide feedback about adherence and offer suggestions. The first session includes psychoeducation about PTSD and a treatment rationale prior to general trauma narrative writing instructions, and specific instructions for completing the first writing session, before completing the first writing (30 minutes) session. Participants are instructed to write about the same trauma event at each following session, with an emphasis on delving into their deepest emotions and thoughts, in as much detail as possible, about the event. All writing sessions begin with specific instructions from the therapist followed by 30 minutes of writing by the participant.
  Interventions: Behavioral: Written Exposure Therapy
- Neutral Topic Writing (Active Comparator): Treatment As Usual (TAU) augmented by a neutral topic writing condition. The neutral topic writing condition involves writing about an assigned topic during each of the five writing sessions. As opposed to writing about trauma, the specific focus of this condition is on writing for 30 minutes about topics related to their life without writing about emotions or opinions. Rather, they are asked to write about specific objects or events in detail, as accurately as possible, and with as much description as possible. All writing sessions begin with specific instructions from the therapist followed by 30 minutes of writing by the participant.
  Interventions: Behavioral: Neutral Topic Writing

INTERVENTIONS:
Behavioral: Written Exposure Therapy — Written Exposure Therapy is a 5 session treatment in which individuals write about their trauma event in a specified manner.
  Other Names: Trauma-focused Treatment
  Arms: Written Exposure Therapy
Behavioral: Neutral Topic Writing — Treatment as Usual augmented by 5 sessions of Neutral Topic Writing which involves writing about specific objects (e.g., what they have eaten over the past week) or events (e.g., what they did since yesterday) in detail without discussing thoughts or feelings.
  Other Names: Control Writing
  Arms: Neutral Topic Writing

SUMMARY:
The proposed project will evaluate the efficacy of written exposure therapy (WET) among Veterans engaged in substance use disorder (SUD) treatment, who present with co-occurring posttraumatic stress disorder (PTSD). While SUD treatment programs traditionally do not address PTSD, effective trauma treatments have been used successfully among those with substance use comorbidities. WET is a brief trauma-focused intervention shown to effectively treat PTSD. In a recent acceptability and feasibility pilot study among Veterans with co-occurring SUD and PTSD, results showed a decrease in PTSD symptoms among participants receiving WET. The goal of the present study is to improve outcomes for Veterans who present for SUD treatment with comorbid SUD/PTSD.

DETAILED DESCRIPTION:
This study is a randomized clinical trial within a Substance Use Disorder (SUD) specialty clinic to evaluate whether treatment as usual (TAU) plus Written Exposure Therapy (WET) is superior to TAU augmented by a neutral topic writing condition on both PTSD and addiction outcomes for Veterans in SUD treatment. Veterans with a current diagnosis of SUD and comorbid PTSD will be randomized to either WET plus TAU or TAU augmented by a neutral topic writing condition. During the first writing session, participants will be asked to write about either a personal traumatic experience (WET) or a neutral topic (control). In sessions 2 through 5, participants will again meet with the study therapist for 45 minutes (maintaining the same writing condition as assigned in session one). Measures of trauma symptoms, distress, and mood will be collected at each writing session, with additional assessments at baseline, at post-treatment (following 5 writing sessions), 8-weeks, and 12-weeks post-baseline assessment. The primary aim of this study is to examine whether WET augmentation of TAU improves trauma symptoms for Veterans with SUD and PTSD who are receiving outpatient SUD treatment compared to TAU with a neutral writing control. The secondary aim will examine whether WET improves SUD outcomes for Veterans with comorbid PTSD compared to TAU with a neutral writing control. If results prove promising, they will support WET as an effective brief, cost efficient, easy to disseminate, adjunct to current SUD treatment for Veterans with comorbid PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veterans ages 18 years old or older;
* Meets DSM-5 criteria for at least one substance use disorder (SUD);
* Meets DSM-5 criteria for PTSD;
* Approved for SUD treatment at VA Connecticut Healthcare System.

Exclusion Criteria:

* Veterans who meet current criteria for schizophrenia, schizophrenia-type disorders, or unmedicated mania or bipolar disorder as determined by QuickSCID-5;
* current suicidal or homicidal risks necessitating a higher level of care;
* Veterans who have received an Evidence-Based Psychotherapy for PTSD protocol within the past 6 months;
* Problems that would prevent a participant from completing the writing intervention or study assessments (e.g., illiteracy). To assess for literacy, participants will read parts of the consent out loud.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | 8-week Post-Baseline Follow-up
  PTSD Checklist for DSM-5 (PCL-5) will be used to collect information on PTSD symptoms. The PCL-5 for DSM-5 is a 20-item self-report measure, selected for its dimensional sensitivity, with higher scores reflecting greater PTSD severity. Scoring is based on how much the patient has been bothered by the symptoms on a scale from "0 = not at all" to "4 = extremely." PCL scores will be collected based upon symptoms experienced in the past month at Baseline as well as each Post-Baseline Follow-up (8-weeks and 12-weeks), while the weekly PCL-5 will be administered at each of the five writing sessions and post-treatment (after 5 writing sessions) assessment. PCL-5 total symptom severity scores range from 0 to 80 with higher scores indicating greater PTSD severity.
PTSD Checklist for DSM-5 (PCL-5) | 12-week Post-Baseline Follow-up
  PTSD Checklist for DSM-5 (PCL-5) will be used to collect information on PTSD symptoms. The PCL-5 for DSM-5 is a 20-item self-report measure, selected for its dimensional sensitivity, with higher scores reflecting greater PTSD severity. Scoring is based on how much the patient has been bothered by the symptoms on a scale from "0 = not at all" to "4 = extremely." PCL scores will be collected based upon symptoms experienced in the past month at Baseline as well as each Post-Baseline Follow-up (8-weeks and 12-weeks), while the weekly PCL-5 will be administered at each of the five writing sessions and post-treatment (after 5 writing sessions) assessment. PCL-5 total symptom severity scores range from 0 to 80 with higher scores indicating greater PTSD severity.

SECONDARY OUTCOMES:
Timeline Follow-Back (TLFB) | 8-week Post-Baseline Follow-up
  Timeline Follow-Back (TLFB) will be provided at baseline, and at post-treatment (after 5 writing sessions), 8-week, and 12-week post-baseline follow-up. Calendar-based interviews using the Timeline Follow-Back (TLFB) method will document the frequency of drug and alcohol use for the 3 months prior to baseline assessment, and during the writing sessions (taken at post-treatment follow-up), 8-week, and 12-week post-baseline follow-up. Following baseline, the TLFB will capture days since last assessment (e.g., days between baseline and post-treatment, post-treatment, and 8-weeks, and 8- to 12-week follow-up). Higher numbers of days of use will equal higher substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Meshberg-Cohen, PhD MS BS, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, anonymized dataset will be created. This dataset may be shared with other investigators, upon written request, under a data use agreement prohibiting the recipient from identifying or re-de-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. The data sharing agreement will also restrict redistribution to third parties and proper acknowledgment of the data source. These datasets will be shared per guidelines provided by VACHS Information Security Officer.
Supporting Information: Study Protocol, SAP
Time Frame: After study completion
Access Criteria: After study completion for no less than 7 years

REFERENCES:
- [Derived] Meshberg-Cohen S, Cook JM, Bin-Mahfouz A, Petrakis IL. Written exposure therapy for veterans with co-occurring substance use disorders and PTSD: Study design of a randomized clinical trial. Contemp Clin Trials. 2024 Apr;139:107475. doi: 10.1016/j.cct.2024.107475. Epub 2024 Feb 15. PMID 38365173